CLINICAL TRIAL: NCT02697032
Title: FDHT-PET to Visualize the Effect on the Androgen Receptor Level by Bicalutamide
Brief Title: FDHT PET and Bicalutamide in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, Principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL2015.0704
Record Dates: First submitted 2015-08-25; First posted 2016-03-03 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: FDHT; PET; Breast cancer; Bicalutamide
MeSH Terms: conditions — Breast Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): At day 0 before start with bicalutamide, a FDHT-PET/CT will be performed, and one after 6 weeks (i.e. 2 weeks after steady-state). The second FDHT-PET will be performed to determine if this scan can be used as a biomarker for early response. Patients will be treated with bicalutamide until progression or unacceptable toxicity is encountered.
  Interventions: Drug: Bicalutamide; Procedure: FDHT PET

INTERVENTIONS:
Drug: Bicalutamide — 150mg
  Other Names: casodex
Procedure: FDHT PET — PET scan
  Other Names: 18F-FDHT PET

SUMMARY:
Rationale: The purpose is to evaluate whether non-invasive in vivo imaging of androgen receptor (AR) presence in metastatic breast cancer patients by means of 18F-fluoro-dihydrotestosterone positron emission tomography (FDHT-PET) can be used to predict (early) treatment response to, and optimal dosing of, the anti androgen bicalutamide. The ultimate goal is to contribute to optimal selection of breast cancer patients for anti androgen treatment. Objective: Feasibility to detect a diffrence in uptake on 18F-FDHT scan after 6 weeks of treatment with bicalutamide in metastatic breast cancer patients. Secondary Objectives: to describe whether changes in 18F-FDHT tracer uptake after six weeks associates with response to bicalutamide, to describe whether changes in AR availability are different for breast cancer subgroups during treatment with bicalutamide and to describe whether 18F-FDHT tracer uptake is influenced by the amount of AR tumor expression. Study design: This is a single arm, one stage feasibility study, which will be executed in the University Medical Center Groningen, The Netherlands. The primary endpoint of the study is to evaluate the difference in 18F-FDHT uptake in tumor lesions after 6 weeks of bicalutamide treatment in patients with AR-positive metastatic breast cancer. Patients will be treated with bicalutamide until progression or unacceptable toxicity is encountered. Study population: The investigators will include 20 postmenopausal metastatic breast cancer patients with an AR positive, HER2 negative tumor. Patients should be restaged clinically with bone scintigraphy and CT scan within a 6 week timeframe of the PET examinations. Intervention: All patients will receive a baseline FDHT-PET scan and start with bicalutamide treatment 150mg daily. During follow-up patients will receive one FDHT-PET scan after 6 weeks. Treatment with bicalutamide will continue until progression or unacceptable toxicity is encountered. Main study endpoint: The percent difference in 18F-FDHT uptake in tumor lesions after 6 weeks of monotherapy bicalutamide. A minimum decrease of 20% in 18F-FDHT uptake after 6 weeks compared to baseline uptake with an α of 0.05 and a power of 80%, is considered clinical significant.

ELIGIBILITY:
Inclusion Criteria:

1. A history of histological proven AR-positive (i.e. >10% staining), HER2-negative metastatic breast cancer (preferably assessment on fresh metastasis biopsy, alternatively archival metastasis biopsy)
2. Tumor progression after at least one line of systemic treatment
3. Measurable disease according to RECIST 1.1; or evaluable disease
4. Age ≥ 18 years
5. Postmenopausal status defined as one of the following:

   * Age ≥60 years
   * Previous bilateral oophorectomy
   * Age <60 years and amenorrhea for >12 months in the absence of interfering hormonal therapies (such as LH-RH agonists and ER-antagonists
   * Age <60 years using ER antagonists should have amenorrhea for >12 months and FSH >24U/L and LH>14U/L
6. Adequate hematological, renal and liver function as follows:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelet count >100 x 109/L
   * White blood cell count >3 x 109/L
   * AST and ALT <3.0 x upper limit of normal (ULN)
   * Alkaline phosphatase <2.5 x ULN
   * Creatinine clearance >50mL/min
   * Lipase/amylase <1/5 x ULN
   * Protrombin time, partial tromboplastin time and INR <1.5 x ULN
7. Written informed consent

Exclusion Criteria:

1. Unable to comply with the protocol
2. Evidence of central nervous metastases
3. Presence of life-threatening visceral metastases
4. Corrected QT interval (QTc) >500millliseconds at screening
5. Recent history of cardiac disease, including myocardial infarction, unstable angina pectoris or uncontrolled arrhythmia within 6 months prior to screening; or evidence of severe congestive heart failure with New York Heart Association severity classification > class I.
6. Recent history of trombo-embolic events within 6 months prior to screening
7. Hepatic impairment (Child-Pugh Class B or C)
8. Severe concurrent disease, infection, co morbid condition that, in the judgment of the investigator would make the patient inappropriate for enrollment
9. The concomitant use of strong CYP3A4 inhibitors (see table 1)
10. Previous anti-androgen treatment
11. Concurrent use of ER-directed anti hormonal therapies
12. Radiotherapy or major surgery within 4 weeks before baseline PET scanning

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
quantify residual AR binding sites in metastatic breast cancer | 6 weeks
  To quantify residual AR binding sites in metastatic breast cancer after 6 weeks of treatment with bicalutamide.

SECONDARY OUTCOMES:
determine whether changes in 18F-FDHT uptake | 6 weeks
  To determine whether changes in 18F-FDHT uptake after 6 weeks associates with response to bicalutamide.
Influence amount of AR tumor expression | 6 weeks
  To determine whether 18F-FDHT tracer uptake is influenced by the amount of AR tumor expression.
Difference in changes in AR availability | 6 weeks
  To determine whether changes in AR availability are different for breast cancer subgroups during treatment with bicalutamide

CONTACTS AND LOCATIONS:
Overall Officials: Carolien P. Schröder, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boers J, Venema CM, de Vries EFJ, Hospers GAP, Boersma HH, Rikhof B, Dorbritz C, Glaudemans AWJM, Schroder CP. Serial [18F]-FDHT-PET to predict bicalutamide efficacy in patients with androgen receptor positive metastatic breast cancer. Eur J Cancer. 2021 Feb;144:151-161. doi: 10.1016/j.ejca.2020.11.008. Epub 2020 Dec 18. PMID 33341447